CLINICAL TRIAL: NCT00887185
Title: Validation/Dissemination Of A Temporal Bone Dissection Simulator
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gregory Wiet (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Gregory Wiet, Clinical Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2006H0194; 5R01DC006458-05 (NIH); NIH Grant 5R01DC006458-05
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Computer Simulation; Education
Keywords: Surgical Simulation; Surgical skills training; Temporal bone surgery; Computer simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Traditional training (Active Comparator): Temporal bone dissection training in cadaveric laboratory. Subjects are provided 2 cadaveric temporal bones and asked to spend 2 weeks practicing the surgical technique of complete mastoidectomy with facial recess approach.
  Interventions: Other: Simulator training for temporal bone surgery
- 2 Simulator training (Experimental): Subjects perform temporal bone surgical dissection training on a simulator.
  Interventions: Other: Simulator training for temporal bone surgery

INTERVENTIONS:
Other: Simulator training for temporal bone surgery — Subjects in experimental arm are asked to spend 2 weeks practicing temporal bone surgical procedures using a computer simulation.
  Other Names: Simulator training; Surgical training

SUMMARY:
Designed to test the efficacy of a computer based virtual simulation for teaching ear surgery.

DETAILED DESCRIPTION:
This research is designed to test the efficacy of a computer based virtual simulation for teaching ear surgery. Subjects will be randomized to training in the usual fashion and training in the simulation environment. Subjects performance will be tested in a standard fashion by dissecting cadaveric temporal bones (human ears) before and after training. The subjects will also perform a dissection in the virtual environment before and after training. The results will be tabulated to compare the different training arms. There is minimal risk associated with the projects and is limited to exposure to cadaveric material. Current training techniques utilize cadaveric material so exposure to this type of material is already a part of the standard training process and this study should not constitute an increased risk beyond what is encountered during their regular training. Demographic information will be obtained for each of the study subject on age, sex, information regarding previous otologic training, year of training and prior experience using computers. The anticipated benefits to society will be that future otologic surgeons can obtain operative experience in a controlled and non threatening environment. They will have access to a greater number of variations in pathology. This will allow each novice surgeon to obtain significantly more experience outside the operating room prior to working with live patients. This will result in less risk to the patient and better trained ear surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in residency for ear, nose and throat training or medical student interested in ear, nose and throat training.

Exclusion Criteria:

* Not enrolled in ENT training program or interest in ENT training.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Performance on temporal bone dissection. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Wiet, MD, Principal Investigator — The Ohio State University, Nationwide Children's Hospital
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Wiet GJ, Schmalbrock P, Powell K, Stredney D. Use of ultra-high-resolution data for temporal bone dissection simulation. Otolaryngol Head Neck Surg. 2005 Dec;133(6):911-5. doi: 10.1016/j.otohns.2005.05.655. PMID 16360513
- [Background] Stredney D, Wiet GJ, Bryan J, Sessanna D, Murakami J, Schmalbrock P, Powell K, Welling B. Temporal bone dissection simulation--an update. Stud Health Technol Inform. 2002;85:507-13. PMID 15458142
- [Background] Wiet GJ, Stredney D, Sessanna D, Bryan JA, Welling DB, Schmalbrock P. Virtual temporal bone dissection: an interactive surgical simulator. Otolaryngol Head Neck Surg. 2002 Jul;127(1):79-83. doi: 10.1067/mhn.2002.126588. PMID 12161735
- [Result] Fernandez SA, Wiet GJ, Butler NN, Welling B, Jarjoura D. Reliability of surgical skills scores in otolaryngology residents: analysis using generalizability theory. Eval Health Prof. 2008 Dec;31(4):419-36. doi: 10.1177/0163278708324444. Epub 2008 Oct 7. PMID 18842619
- [Result] Butler NN, Wiet GJ. Reliability of the Welling scale (WS1) for rating temporal bone dissection performance. Laryngoscope. 2007 Oct;117(10):1803-8. doi: 10.1097/MLG.0b013e31811edd7a. PMID 17721407